CLINICAL TRIAL: NCT03673501
Title: A Phase 3, Interventional, Randomized, Multicenter, Open-Label Study of Ripretinib vs Sunitinib in Patients With Advanced Gastrointestinal Stromal Tumor (GIST) After Treatment With Imatinib
Brief Title: A Study of Ripretinib vs Sunitinib in Advanced GIST Patients After Treatment With Imatinib
Acronym: INTRIGUE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCC-2618-03-002
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ripretinib (Experimental): Ripretinib (150 mg) once a day continuous dosing for 6-week (42 days) cycles
  Interventions: Drug: Ripretinib
- Sunitinib (Active Comparator): Sunitinib (50 mg) once a day in 6-week (42 days) cycles with 4 weeks continuous dosing followed by 2 week break.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Ripretinib — Oral KIT/PDGFRA kinase inhibitor
  Other Names: DCC-2618
  Arms: Ripretinib
Drug: Sunitinib — Oral receptor tyrosine kinase (RTK) inhibitor
  Other Names: Sutent
  Arms: Sunitinib

SUMMARY:
This is a 2-arm, randomized, open-label, international, multicenter study comparing the efficacy of ripretinib to sunitinib in GIST patients who progressed on or were intolerant to first-line anticancer treatment with imatinib. Approximately 426 patients will be randomized in a 1:1 ratio to ripretinib 150 mg once daily (continuous dosing for 6 week cycles) or sunitinib 50 mg once daily (6 week cycles, 4 weeks on, 2 weeks off).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age at the time of informed consent.
2. Histologic diagnosis of GIST and must be able to provide an archival tumor tissue sample, otherwise, a fresh biopsy is required.
3. Molecular pathology report must be available. If molecular pathology report is not available or insufficient, an archival tumor tissue sample or fresh biopsy is required for mutation status confirmation by the central laboratory prior to randomization.
4. Patients must have progressed on imatinib or have documented intolerance to imatinib.
5. Eastern Cooperative Oncology Group (ECOG) Performance Score (PS) of ≤ 2 at screening.
6. Female patients of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test at screening and negative pregnancy test at Cycle 1 Day 1 prior to the first dose of study drug.
7. Patients of reproductive potential must agree to follow the contraception requirements outlined in the study protocol.
8. Patients must have at least 1 measurable lesion according to Modified Response Evaluation Criteria in Solid Tumors (mRECIST) Version 1.1 (non nodal lesions must be ≥ 1.0 cm in the long axis or ≥ double the slice thickness in the long axis) within 21 days prior to the first dose of study drug.
9. Adequate organ function and bone marrow reserve as indicated by the central laboratory assessments performed at screening.
10. Resolution of all toxicities from prior therapy to ≤ Grade 1 (or patient baseline) within 1 week prior to the first dose of study drug (excluding alopecia and ≤ Grade 3 clinically asymptomatic lipase, amylase, and creatine phosphokinase laboratory abnormalities).
11. The patient is capable of understanding and complying with the protocol and the patient has signed the informed consent document. Signed informed consent form (ICF) must be obtained before any study-specific procedures are performed and the patient must agree to not participate in any other interventional clinical trial while on treatment in this clinical trial. Participation in a noninterventional study (including observational studies) is permitted.

Exclusion Criteria:

1. Treatment with any other line of therapy in addition to imatinib for advanced GIST. Imatinib-containing combination therapy in the first-line setting is not allowed.
2. Patients with a prior or concurrent malignancy whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of this clinical trial are not eligible.
3. Patient has known active central nervous system metastases.
4. New York Heart Association class II-IV heart disease, myocardial infarction within 6 months of cycle 1 day 1, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension or congestive heart failure.
5. Left ventricular ejection fraction (LVEF) < 50% at screening.
6. Arterial thrombotic or embolic events such as cerebrovascular accident (including ischemic attacks) or hemoptysis within 6 months before the first dose of study drug.
7. Venous thrombotic events (e.g. deep vein thrombosis) or pulmonary arterial events (e.g. pulmonary embolism) within 1 month before the first dose of study drug. Patients on stable anticoagulation therapy for at least one month are eligible.
8. 12-lead ECG demonstrating QT interval corrected (QTc) by Fridericia's formula > 450 ms in males or > 470 ms in females at screening or history of long QTc syndrome
9. Use of known substrates or inhibitors of breast cancer resistance protein (BCRP) transporters within 14 days or 5 x the half-life (whichever is longer) prior to the first dose of study drug.
10. Major surgeries (e.g. abdominal laparotomy) within 4 weeks of the first dose of study drug. All major surgical wounds must be healed and free of infection or dehiscence before the first dose of study drug.
11. Any other clinically significant comorbidities.
12. Known human immunodeficiency virus or hepatitis C infection only if the patient is taking medications that are excluded per protocol, active hepatitis B, or active hepatitis C infection.
13. If female, the patient is pregnant or lactating.
14. Known allergy or hypersensitivity to any component of the study drug.
15. Gastrointestinal abnormalities including but not limited to:

    * inability to take oral medication
    * malabsorption syndromes
    * requirement for intravenous (IV) alimentation
16. Any active bleeding excluding hemorrhoidal or gum bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (120):
- United States (43):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of California San Diego Medical Center, La Jolla, California
  - UCLA Hematology Oncology Center - Main Site, Los Angeles, California
  - Stanford Medicine, Stanford, California
  - University of Colorado Hospital - Anschutz Cancer Pavillion, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Smilow Cancer Hospital at Yale, New Haven, Connecticut
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic Florida, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Orlando Health UF Health Cancer Center, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Georgia Cancer Specialists, Sandy Springs, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - IU Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Norton Cancer Institute, Audubon Hospital Campus, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Monter Cancer Center, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center-Montefiore Medical Park, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Comprehensive Cancer Center - Arthur G. James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - University of Toledo, Toledo, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University Center for Health and Healing, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Froedtert Hospital-Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (2):
  - Sanatorio Allende, Córdoba, Córdoba Province
  - Instituto Medicao Especializado Alexander Fleming, Buenos Aires
- Australia (6):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Princess Alexandara Hospital, Woolloongabba
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - UZ Leuven, Leuven
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Québec
- Clinica San Carlos de Apoquindo Red Salud UC Christs, Santiago, Chile
- Fakultni nemocnice v Motole, Prague, Czechia
- France (9):
  - Institut Bergonnié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hopital La Timone, Marseille
  - IPC, Marseille
  - IGR, Paris
  - CHU Poitiers-Hopital la Miletrie, Poitiers
  - ICO - Site René Gauducheau, Saint-Herblain
- Germany (3):
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Technische Universitat Dresden, Dresden
  - West German Cancer Center, Essen
- Hungary (2):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Debreceni Egyetem, Debrecen
- Israel (3):
  - Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov
  - Rabin Medical Cente, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - stituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Universita degli Studi di Palermo, Palermo
  - Università Campus Bio-Medico di Roma, Rome
- Netherlands (4):
  - Antoni van Leeuwenhoek, Amsterdam
  - The Netherlands Cancer Institute, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Centre, Leiden
- Oslo University Hospital, Oslo, Norway
- Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw, Poland
- National Cancer Centre, Singapore, Singapore
- South Korea (4):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (12):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario HM Madrid Sanchinarro, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano de Oncología,, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
- Karolinska universitetssjukhuset, Solna, Sweden
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Fondation du Centre Pluridisciplinaire d'Oncologi, Lausanne
  - Universitaetsspital Zuerich, Klinik fuer Onkologie, Zurich
- Taiwan (5):
  - Chang Gung Memorial Hospital, Linkou District, Taoyuan County
  - Kaohsiung Chang Gung Memorial Hospital,, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Chen Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (5):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's University Hospital, Leeds
  - Royal Marsden Hospital - Fulham, London
  - University College London Hospitals, London
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heinrich MC, Blay JY, Gelderblom H, George S, Schoffski P, von Mehren M, Zalcberg JR, Jones RL, Kang YK, Razak AA, Trent J, Attia S, Le Cesne A, Boye K, Goldstein D, Sanchez C, Siontis BL, Cox P, Davis E, Sherman ML, Ruiz-Soto R, Bauer S. Updated Overall Survival and Long-Term Safety With Ripretinib Versus Sunitinib in Patients With GI Stromal Tumor: Final Overall Survival Analysis From INTRIGUE. J Clin Oncol. 2025 Jul 10;43(20):2239-2244. doi: 10.1200/JCO-24-02818. Epub 2025 May 23. PMID 40408605
- [Derived] Heinrich MC, Jones RL, George S, Gelderblom H, Schoffski P, von Mehren M, Zalcberg JR, Kang YK, Razak AA, Trent J, Attia S, Le Cesne A, Siontis BL, Goldstein D, Boye K, Sanchez C, Steeghs N, Rutkowski P, Druta M, Serrano C, Somaiah N, Chi P, Reichmann W, Sprott K, Achour H, Sherman ML, Ruiz-Soto R, Blay JY, Bauer S. Ripretinib versus sunitinib in gastrointestinal stromal tumor: ctDNA biomarker analysis of the phase 3 INTRIGUE trial. Nat Med. 2024 Feb;30(2):498-506. doi: 10.1038/s41591-023-02734-5. Epub 2024 Jan 5. PMID 38182785
- [Derived] Gelderblom H, Jones RL, Blay JY, George S, von Mehren M, Zalcberg JR, Kang YK, Razak AA, Trent J, Attia S, Le Cesne A, Siontis BL, Goldstein D, Boye K, Sanchez C, Steeghs N, Rutkowski P, Druta M, Serrano C, Somaiah N, Chi P, Harrow B, Becker C, Reichmann W, Sherman ML, Ruiz-Soto R, Heinrich MC, Bauer S; INTRIGUE investigators. Patient-reported outcomes and tolerability in patients receiving ripretinib versus sunitinib after treatment with imatinib in INTRIGUE, a phase 3, open-label study. Eur J Cancer. 2023 Oct;192:113245. doi: 10.1016/j.ejca.2023.113245. Epub 2023 Jul 20. PMID 37598656
- [Derived] Bauer S, Jones RL, Blay JY, Gelderblom H, George S, Schoffski P, von Mehren M, Zalcberg JR, Kang YK, Razak AA, Trent J, Attia S, Le Cesne A, Su Y, Meade J, Wang T, Sherman ML, Ruiz-Soto R, Heinrich MC. Ripretinib Versus Sunitinib in Patients With Advanced Gastrointestinal Stromal Tumor After Treatment With Imatinib (INTRIGUE): A Randomized, Open-Label, Phase III Trial. J Clin Oncol. 2022 Dec 1;40(34):3918-3928. doi: 10.1200/JCO.22.00294. Epub 2022 Aug 10. PMID 35947817
- [Derived] Nemunaitis J, Bauer S, Blay JY, Choucair K, Gelderblom H, George S, Schoffski P, Mehren MV, Zalcberg J, Achour H, Ruiz-Soto R, Heinrich MC. Intrigue: Phase III study of ripretinib versus sunitinib in advanced gastrointestinal stromal tumor after imatinib. Future Oncol. 2020 Jan;16(1):4251-4264. doi: 10.2217/fon-2019-0633. Epub 2019 Nov 22. PMID 31755321
- See also: Deciphera Company Website — http://www.deciphera.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ripretinib | Sunitinib
Started | 226 | 227
Completed (Completed patients are defined as patients that are followed until death or until the sponsor terminates the study.) | 190 | 203
Not Completed | 36 | 24
Not completed — Participants ongoing. | 36 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ripretinib | Sunitinib | Total
Number analyzed (Participants) | 226 | 227 | 453
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 145 | 143 | 288
  65-74 years | 56 | 66 | 122
  75 years and older | 25 | 18 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 85 | 172
  Male | 139 | 142 | 281
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 14 | 14 | 28
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 31 | 27 | 58
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  White | 148 | 152 | 300
  Not Report | 30 | 30 | 60
  Other | 1 | 2 | 3
Eastern Cooperative Oncology Group (ECOG) Score at Screening [Count of Participants; unit: Participants] — An ECOG Score of 0 means the participant is fully active, able to carry on all pre-disease performance without restriction
  ECOG Score of 1 means the participant is restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work
  ECOG Score of 2 means the participant is ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    ECOG Score 0 | 131 | 128 | 259
    ECOG Score 1 | 92 | 98 | 190
    ECOG Score 2 | 3 | 1 | 4
Mutation Type per Electronic Data Capture (EDC) [Count of Participants; unit: Participants] — Electronic Data Capture (EDC) is a system used to capture patient information in a clinical trial. The data is presented based on how many participants had the KIT proto-oncogene receptor tyrosine kinase (KIT) Exon 9 mutation, KIT Exon 11 mutation, the KIT/platelet-derived growth factor receptor alpha (PDGFRA) wild type (WT) mutation, or other KIT (absence of Exon 9 or 11)/PDGFRA mutations.
  Participants
    KIT Exon 9 | 31 | 28 | 59
    KIT Exon 11 | 167 | 169 | 336
    KIT/PDGFRA WT | 14 | 16 | 30
    Other KIT (absence of Exon 9 or 11)/PDGFRA | 14 | 14 | 28
Intolerance to Imatinib per Electronic Data Capture (EDC) [Count of Participants; unit: Participants] — Electronic Data Capture (EDC) is a system used to capture patient information in a clinical trial. The data is presented based on participants that were intolerant to imatinib or not.
  Participants
    Yes | 15 | 19 | 34
    No | 211 | 208 | 419
Mutation Type per Interactive Response Technology (IRT) [Count of Participants; unit: Participants] — Interactive Response Technology (IRT) is a randomization and trial supply system that randomly assigns patients to one of the study treatments and supplies study drug. The data is presented based on the participant's Mutational Status: KIT exon 9 mutation; KIT exon 11 mutation; KIT/PDGFRA wild type (WT); or other KIT (absence of exon 9 or 11)/PDGFRA mutations
  Participants
    KIT Exon 9 | 31 | 29 | 60
    KIT Exon 11 | 163 | 164 | 327
    KIT/PDGFRA wild type (WT) | 15 | 18 | 33
    Other KIT (absence of Exon 9 or 11)/PDGFRA | 17 | 16 | 33
Intolerance to Imatinib per Interactive Response Technology (IRT) [Count of Participants; unit: Participants] — Interactive Response Technology (IRT) is a randomization and trial supply system that randomly assigns patients to one of the study treatments and supplies study drug. The data is presented based on whether the participants were intolerant to imatinib or not.
  Participants
    Yes | 22 | 23 | 45
    No | 204 | 204 | 408

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) in the KIT Exon 11 Intent to Treat (ITT) Population
Description: PFS is defined as the interval between the date of randomization and the earliest documented evidence of disease progression based on the independent radiologic review using modified RECIST Version 1.1-(mRECIST 1.1) GIST specific, or death due to any cause. Per mRECIST 1.1, progression was defined using mRECIST 1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From date of randomization to earliest documented evidence of disease progression, or death due to any cause (up to 2.1 years)
Population: The KIT Exon 11 Intent to Treat (ITT) Population is defined as all patients who are designated as having a mutation in KIT Exon 11 at the time of randomization. Patients in this population will be analyzed according to the treatment they were scheduled to receive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ripretinib | Sunitinib
Number analyzed (Participants) | 163 | 164
months | 8.3 [6.8 to 13.3] | 7.0 [5.6 to 10.9]
Statistical Analysis 1: Comparison: Ripretinib vs Sunitinib; Test type: Superiority; p = 0.3598, Log Rank; Strata: by intolerance to imatinib treatment; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.66 to 1.16]

2. Primary Outcome: Progression Free Survival (PFS) in the All Patient (AP) Intent to Treat (ITT) Population
Description: PFS is defined as the interval between the date of randomization and the earliest documented evidence of disease progression based on the independent radiologic review using modified RECIST Version 1.1-(mRECIST 1.1) Gastrointestinal stromal tumor (GIST) specific, or death due to any cause. Per mRECIST 1.1, progression was defined using mRECIST 1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: as for outcome 1
Population: All patient (AP) Intent to Treat (ITT) Population is defined as all patients who are randomized. Patients in this population will be analyzed according to the treatment they were scheduled to receive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ripretinib | Sunitinib
Number analyzed (Participants) | 226 | 227
months | 8.0 [6.5 to 10.8] | 8.3 [6.3 to 11.0]
Statistical Analysis 1: Comparison: Ripretinib vs Sunitinib; Test type: Superiority; p = 0.7153, Log Rank — Two-sided P-value; Strata: mutation status (KIT exon 9 vs. 11 vs. KIT/PDGFRA WT vs. other KIT {absence of exon 9 or 11}/PDGFRA) and intolerance to imatinib treatment; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.82 to 1.33]

3. Secondary Outcome: Objective Response Rate (ORR) in the KIT Exon 11 Intent to Treat (ITT) Population Population
Description: ORR was defined as the proportion of patients with confirmed complete response (CR) + confirmed partial response (PR) based on independent radiologic review using modified RECIST (mRECIST) criteria as best overall response. Per mRECIST 1.1 criteria, complete response is defined as disappearance of all target lesions; partial response is defined as >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: From confirmed CR or PR to disease progression (up to 1.74 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ripretinib | Sunitinib
Number analyzed (Participants) | 163 | 164
percentage of participants | 23.9 [17.6 to 31.2] | 14.6 [9.6 to 21.0]
Statistical Analysis 1: Comparison: Ripretinib vs Sunitinib; Test type: Superiority; p = 0.0333, Cochran-Mantel-Haenszel; Strata: intolerance to imatinib treatment

4. Secondary Outcome: Objective Response Rate (ORR) in the All Patient (AP) Intent to Treat (ITT) Population
Description: as for outcome 3
Time Frame: From confirmed CR or PR to disease progression (up to 1.74 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ripretinib | Sunitinib
Number analyzed (Participants) | 226 | 227
percentage of participants | 21.7 [16.5 to 27.6] | 17.6 [12.9 to 23.2]
Statistical Analysis 1: Comparison: Ripretinib vs Sunitinib; Test type: Superiority; p = 0.2681, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Overall Survival (OS) in the KIT Exon 11 Intent to Treat (ITT) Population
Description: OS was defined as the time from the date of randomization until death due to any cause.
Time Frame: From date of randomization until death due to any cause (up to 3.33 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ripretinib | Sunitinib
Number analyzed (Participants) | 163 | 164
months | 34.0 [29.3 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to fewer number of participants with events | 31.5 [29.4 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to fewer number of participants with events
Statistical Analysis 1: Comparison: Ripretinib vs Sunitinib; Test type: Superiority; p = 0.7733, Log Rank; Strata: intolerance to imatinib treatment; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.75 to 1.48]

6. Secondary Outcome: Overall Survival (OS) in the All Patient (AP) Intent to Treat (ITT) Population
Description: OS was defined as the time from the date of randomization until death due to any cause.
Time Frame: From date of randomization until death due to any cause (up to 3.33 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ripretinib | Sunitinib
Number analyzed (Participants) | 226 | 227
months | 35.5 [29.3 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to fewer number of participants with events | 30.9 [28.9 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to fewer number of participants with events
Statistical Analysis 1: Comparison: Ripretinib vs Sunitinib; Test type: Superiority; p = 0.3928, Log Rank; Strata: mutation status (KIT exon 9 vs. 11 vs. KIT/PDGFRA WT vs. other KIT {absence of exon 9 or 11}/PDGFRA) and intolerance to imatinib; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.66 to 1.18]

ADVERSE EVENTS:
Time Frame: Collection of Adverse events started from the signing of informed consent through safety follow-up (up to 3.22 years)
Description: The Safety Population is defined as all patients who are randomized and receive at least one dose of study drug.
Arm/Group | Ripretinib | Sunitinib
All-Cause Mortality (participants affected / at risk) | 90/223 | 95/221
Serious Adverse Events (participants affected / at risk) | 64/223 | 61/221
Other Adverse Events (participants affected / at risk) | 221/223 | 219/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ripretinib (N=223) | Sunitinib (N=221)
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 6
Ascites (Gastrointestinal disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemoperitoneum (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 5 | 0
Localised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 5 | 2
Cellulitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 3
Abdominal abscess (Infections and infestations) | 1 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Anorectal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
Escherichia peritonitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 1
Psychomotor retardation (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 2
Hypertensive urgency (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Supraventricular extrasustoles (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Acquired encephalocele (Injury, poisoning and procedural complications) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ripretinib (N=223) | Sunitinib (N=221)
Anaemia (Blood and lymphatic system disorders) | 25 | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 14
Neutropenia (Blood and lymphatic system disorders) | 0 | 28
Constipation (Gastrointestinal disorders) | 79 | 48
Abdominal pain (Gastrointestinal disorders) | 57 | 35
Nausea (Gastrointestinal disorders) | 54 | 56
Diarrhoea (Gastrointestinal disorders) | 47 | 107
Vomiting (Gastrointestinal disorders) | 27 | 31
Dyspepsia (Gastrointestinal disorders) | 19 | 38
Abdominal distension (Gastrointestinal disorders) | 17 | 16
Stomatitis (Gastrointestinal disorders) | 18 | 81
Abdominal pain upper (Gastrointestinal disorders) | 13 | 23
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 35
Dry mouth (Gastrointestinal disorders) | 6 | 13
Oral pain (Gastrointestinal disorders) | 3 | 13
Fatigue (General disorders) | 84 | 91
Asthenia (General disorders) | 38 | 41
Oedema peripheral (General disorders) | 19 | 21
Pyrexia (General disorders) | 14 | 20
Weight decreased (Investigations) | 40 | 29
Blood bilirubin increased (Investigations) | 20 | 16
Lipase increased (Investigations) | 19 | 20
Aspartate aminotransferase increased (Investigations) | 15 | 24
Alanine aminotransferase increased (Investigations) | 13 | 15
Neutrophil count decreased (Investigations) | 2 | 42
Platelet count decreased (Investigations) | 2 | 32
White blood cell count decreased (Investigations) | 1 | 22
Decreased appetite (Metabolism and nutrition disorders) | 60 | 54
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 11
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 81 | 25
Muscle spasms (Musculoskeletal and connective tissue disorders) | 59 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 36
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 16
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 | 3
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 | 6
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 12
Dizziness (Nervous system disorders) | 15 | 18
Dysgeusia (Nervous system disorders) | 8 | 33
Insomnia (Psychiatric disorders) | 19 | 13
Anxiety (Psychiatric disorders) | 14 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 144 | 18
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 61 | 116
Pruritus (Skin and subcutaneous tissue disorders) | 49 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 33 | 34
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 | 18
Pain of skin (Skin and subcutaneous tissue disorders) | 18 | 5
Rash (Skin and subcutaneous tissue disorders) | 17 | 14
Actinic keratosis (Skin and subcutaneous tissue disorders) | 15 | 5
Hair colour changes (Skin and subcutaneous tissue disorders) | 5 | 11
Hypertension (Vascular disorders) | 60 | 106
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 0
Blood creatine phosphokinase increased (Investigations) | 7 | 11
Headache (Nervous system disorders) | 36 | 39
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT03673501/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT03673501/SAP_001.pdf